CLINICAL TRIAL: NCT01832974
Title: A Phase I/II Trial of IL-13-PE in Patients With Treatment Refractory Malignancies With a Focus on Metastatic and Locally Advanced Adrenocortical Carcinoma
Brief Title: Possible New Therapy for Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision by the sponsor during Phase 1.
Sponsor: INSYS Therapeutics Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-C-0046; 13-C-0046 D (Other: National Institutes of Health Clinical Center); P11946 (Other: INSYS Therapeutics Inc)
Record Dates: First submitted 2012-09-11; First posted 2013-04-16 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenal Gland Cancer; Treatment Refractory Malignancies; Metastatic Cancer
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Gland Neoplasms; Neoplasm Metastasis

ARMS (4):
- Part 1- 1 μg/kg (Other): Up to 6 participants receiving IL-13-PE 1 μg/kg (rounded down to the nearest vial size within 10% of the calculated dose), intravenous (IV), Days 1, 3 and 5 in each monthly cycle for up to 4 cycles
  Interventions: Drug: IL-13-PE
- Part 1 - 2 μg/kg (Other): If lower dose was tolerated, 3-6 participants receiving IL-13-PE 2 μg/kg (rounded down to the nearest vial size within 10% of the calculated dose), intravenous (IV), Days 1, 3 and 5 in each monthly cycle for up to 4 cycles
  Interventions: Drug: IL-13-PE
- Part 1 - 3 μg/kg (Other): If lower dose was tolerated, 3-6 participants receiving IL-13-PE 3 μg/kg (rounded down to the nearest vial size within 10% of the calculated dose), intravenous (IV), Days 1, 3 and 5 in each monthly cycle for up to 4 cycles
  Interventions: Drug: IL-13-PE
- Part 2 - All Participants (Experimental): All participants in Part 2, receiving maximum tolerated dose of IL-13-PE 1-3 μg/kg (rounded down to the nearest vial size within 10% of the calculated dose), intravenous (IV), 3 times per monthly cycle for up to 4 cycles (or longer for participants receiving clinical benefit)
  Interventions: Drug: IL-13-PE

INTERVENTIONS:
Drug: IL-13-PE — IL-13-PE intravenous infusion
  Other Names: Interleukin-13 PE38QQR

SUMMARY:
IL-13-PE is a chemical similar to one made by the body that is connected to a toxin to specifically attack cancer cells. Researchers want to look at different doses of IL-13-PE to find one that may be safe and effective against cancer that has returned, spread to other organs, or that cannot be surgically removed.

Participants will receive physical exams and report side effects. Blood and urine samples will be collected. Imaging studies, tissue samples, and other tests will be used to study the tumor before the start of treatment and during the study. IL-13-PE therapy will be given to each participant on days 1, 3 and 5 of each monthly cycle for up to 4 monthly cycles.

The study will be done in two parts, with a six-month period between them. If the cancer continues to grow, participants will stop taking IL-13-PE. If the cancer continues to shrink or not grow the study will continue, even into a follow-up period after the second part of the study.

The first part of this study will determine how much IL-13-PE can be tolerated. For this part, the study is recruiting adult patients with various types of cancer. After six participants have taken the lowest dose with no more than one experiencing dose-limiting toxicity, two participants may begin the study taking the medium dose. If they tolerate the medium dose for a month, up to four more may begin at that dose. When at least three participants have tolerated the medium dose, two may attempt the highest dose. When they have tolerated the highest dose for one monthly cycle, 1-4 more may begin the study, receiving the highest dose.

Adrenal cortex cancer (ACC) is a rare tumor in the gland above the kidney. It affects only 1-2 people per million each year and causes hormone problems. This tumor affects children under age 5 and adults aged 30-40, causing death within five years for up to 80% of them. During the second part of the study, all participants will be ACC patients. They will receive the highest dose tolerated during Part 1 on days 1, 3, and 5 of each monthly cycle for up to four months.

ELIGIBILITY:
Inclusion Criteria:

* Has measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria at presentation
* Has failed standard treatment
* Has met protocol-specified criteria for qualification and contraception
* Has voluntarily consented to participate and provided written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:
* the safety or well-being of the participant or study staff
* the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
* the analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of IL-13-PE | during 16-week dose-escalation treatment, up to 3 years
Best overall response | during 16-week treatment, up to 3 years

SECONDARY OUTCOMES:
Percentage of participants with clinically significant abnormal findings on physical examination | during 16-week treatment and 12-month follow-up, up to 4 years
Percentage of participants with clinically significant abnormal findings on laboratory evaluation | during 16-week treatment and 12-month follow-up, up to 4 years

OTHER OUTCOMES:
Estimated Progression-Free Survival | during 16-week treatment and 12-month follow-up, up to 4 years
Survival | Indefinitely
  Following the 12-month follow-up evaluation patients will be followed via phone or e-mail contact every 6 months for survival

CONTACTS AND LOCATIONS:
Overall Officials: Electron Kebebew, M.D., Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Cancer Institute at the National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jain M, Zhang L, He M, Patterson EE, Nilubol N, Fojo AT, Joshi B, Puri R, Kebebew E. Interleukin-13 receptor alpha2 is a novel therapeutic target for human adrenocortical carcinoma. Cancer. 2012 Nov 15;118(22):5698-708. doi: 10.1002/cncr.27629. Epub 2012 May 8. PMID 22570059
- [Background] Bilimoria KY, Shen WT, Elaraj D, Bentrem DJ, Winchester DJ, Kebebew E, Sturgeon C. Adrenocortical carcinoma in the United States: treatment utilization and prognostic factors. Cancer. 2008 Dec 1;113(11):3130-6. doi: 10.1002/cncr.23886. PMID 18973179
- [Background] Fassnacht M, Libe R, Kroiss M, Allolio B. Adrenocortical carcinoma: a clinician's update. Nat Rev Endocrinol. 2011 Jun;7(6):323-35. doi: 10.1038/nrendo.2010.235. Epub 2011 Mar 8. PMID 21386792